CLINICAL TRIAL: NCT04381793
Title: Treatment of CFS & Fibromyalgia With Recovery Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Practitioners Alliance Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAN study 2019-10
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-02

CONDITIONS: Fibromyalgia; Chronic Fatigue Syndrome
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic

STUDY DESIGN:
Intervention Model Description: Open pilot study to assess efficacy and antibody effects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessing clinical efficacy (Experimental): Subjects will receive four tablets twice a day (three times a day for five day loading dose), taking the treatment for 5 - 6 weeks. The treatment is a unique nutritional peptide mix derived from porcine serum. Pre-and post FIQ-R and VA symptom score will be assessed as well as overall well-being. In a subgroup, pre-and post antibody levels will also be checked. Phase 1 will be a group of 60 subjects
  Interventions: Dietary Supplement: Recovery Factors

INTERVENTIONS:
Dietary Supplement: Recovery Factors — Porcine serum amino acid/peptide

SUMMARY:
The study will explore if Recovery Factors improve symptoms in fibromyalgia and chronic fatigue syndrome

DETAILED DESCRIPTION:
Subjects will receive four tablets twice a day (three times a day for five day loading dose), taking the treatment for 5 - 6 weeks. Subjects will receive four tablets twice a day (three times a day for five day loading dose), taking the treatment for 5 - 6 weeks. The treatment is a unique nutritional peptide mix derived from porcine serum

ELIGIBILITY:
Inclusion Criteria:

* Meet ACR 2010 amended Fibromyalgia criteria or CDC CFS Criteria Overall well being score of 5 of less (on 0-10 VAS)

Exclusion Criteria:

Pregnant Clotting disorders

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-07-04 (Actual); Study Completion 2020-07-04 (Actual)

PRIMARY OUTCOMES:
VAS | 6 weeks
  Composite VAS (1-10) for Fatigue, Pain, Cognition, Sleep and overall well-being

SECONDARY OUTCOMES:
antibody titres | 10 weeks
  Total IgG and IgG 1-4 subsets
FIQ-R | 6 weeks
  Fibromyalgia severity scale

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morello, ND, Principal Investigator — Woman's Hospital in Vancouver
Locations (1):
- Jacob Teitelbaum MD, Kailua, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No